CLINICAL TRIAL: NCT02207309
Title: A Randomized, Double Blind, Phase II Trial of Pazopanib Versus Placebo as Maintenance Therapy in Patients With Retroperitoneal and Visceral High-risk Soft Tissue Sarcomas Following Prior Neo- and/or Adjuvant Doxorubicin / Ifosfamide Chemotherapy With Regional Hyperthermia
Brief Title: Pazopanib Maintenance Phase II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Lars Lindner, PD Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NPM001; 2013-000522-58 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Sarcoma
Keywords: high-risk soft tissue sarcoma; pazopanib; retroperitoneal soft tissue sarcoma; visceral soft tissue sarcoma; votrient
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pazopanib (Active Comparator): 800mg, oral, 24 months
  Interventions: Drug: Pazopanib
- Placebo (Placebo Comparator): 800mg, oral, 24 months
  Interventions: Drug: Placebo (for Pazopanib)

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient
  Arms: Pazopanib
Drug: Placebo (for Pazopanib)
  Arms: Placebo

SUMMARY:
This trial compares pazopanib to placebo as maintenance treatment over 2 years in patients with retroperitoneal and visceral high-risk soft tissue sarcomas after multimodal treatment including prior neo- and/or adjuvant doxorubicin / ifosfamide chemotherapy with regional hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up
* Patients must have histological evidence of high-grade soft tissue sarcoma (grade 2 - 3) according to the FNLCC grading system, tumor size ≥ 5 cm and deep localization with regard to the superficial fascia, excluding the following tumor types:

  * Embryonal rhabdomyosarcoma
  * Chondrosarcoma (excluding extraskeletal myxoid chondrosarcoma)
  * Osteosarcoma (excluding extraskeletal osteosarcoma)
  * Ewing tumors / primitive neuroectodermal tumor (PNET)
  * Gastro-intestinal stromal tumors (GIST)
  * Dermatofibrosarcoma protuberans
* Patients who had undergone previous surgery with inadequate margins (tumour-free margins ≤1 cm or margins contaminated) are eligible if thermochemotherapy has been started within 8 weeks after surgery
* Unstained slides and ideally tumour blocks must be available for histological central review
* Completed 4 to 8 cycles of thermochemotherapy with doxorubicin and ifosfamide at least 21 days but no more than 42 days prior to study entry
* No evidence of disease following completion of first-line thermochemotherapy and within ≤ 21 days of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No other prior chemotherapy except thermochemotherapy with doxorubicin and ifosfamide
* Adequate organ system function

Exclusion Criteria:

* No prior or concurrent second primary malignant tumors (except adequately treated in situ carcinoma of cervix, or basal cell carcinoma)
* No symptomatic or known Central nervous system (CNS) metastases at baseline
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel.
* Corrected QT interval (QTc) > 480 msecs
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) (See Appendix D for description)
* Poorly controlled hypertension (SBP of ≤ 150 mmHg or DBP of ≤95 mmHg is acceptable provided that BP will be treated and monitored at least weekly. The goal is to attain controlled hypertension within 4 weeks of start of IMP which is defined as grade ≤1 hypertension CTCAE Version 4.0)
* NYHA II at Screening for Patients > 65 years
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible

* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage Note: Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions).

  * Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.
  * Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
* Recent hemoptysis (≥½ teaspoon of red blood within 8 weeks before first dose of study drug).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Treatment with any of the following anti-cancer therapies:

  * radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lindner, MD, PhD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig-Maximilians University of Munich, Klinikum Großhadern, Munich, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Targeted recruitment goal were 150 patients, 1 patient was randomised
Pre-assignment Details: Contrary to the original expectation, patients with retroperitoneal or visceral high-risk soft tissue sarcoma were generally not prepared to undergo further therapy with pazopanib for 2 years after multimodal therapy consisting of 8 cycles of chemotherapy in combination with hyperthermia, surgery and, if necessary, radiotherapy, which may have side effects.
Groups:
- Pazopanib: 800mg, oral, 24 months
  Pazopanib
- Placebo: 800mg, oral, 24 months
  Placebo (for Pazopanib)
Period: Overall Study
Arm/Group | Pazopanib | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Contrary to the original expectation, patients with high-risk retroperitoneal or visceral soft tissue sarcoma after multimodal therapy consisting of 8 cycles of chemotherapy in combination with hyperthermia, surgery, and possibly radiotherapy were generally unwilling to undergo further therapy with pazopanib over 2 years, which may have had side effects. Hence only 1 participant was recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  Germany | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The study could not be evaluated. Only one patient was included.
Time Frame: Study Start Dat: June 22, 2015; Study Completion Date: July 29, 2016 ; an approximate study duration of 13 months
Population: The study could not be evaluated. Only one patient was included.
  Contrary to the original expectation, patients with retroperitoneal or visceral high-risk soft tissue sarcoma were generally not prepared to undergo further therapy with pazopanib for 2 years after multimodal therapy consisting of 8 cycles of chemotherapy in combination with hyperthermia, surgery and, if necessary, radiotherapy, which may have side effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: The study could not be evaluated. Only one patient was included.
Time Frame: Study Start Dat: June 22, 2015; Study Completion Date: July 29, 2016 ; an approximate study duration of 13 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study Start Dat: June 22, 2015; Study Completion Date: July 29, 2016; an approximate study duration of 13 months
Description: Contrary to the original expectation, patients with high-risk retroperitoneal or visceral soft tissue sarcoma after multimodal therapy consisting of 8 cycles of chemotherapy in combination with hyperthermia, surgery, and possibly radiotherapy were generally unwilling to undergo further therapy with pazopanib over 2 years, which may have had side effects. Hence only 1 participant was recruited.
Arm/Group | Pazopanib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes